CLINICAL TRIAL: NCT01739712
Title: Students With Diabetes: Does Optimizing Sleep Promote Classroom, Behavioral, and Disease-Related Improvement
Brief Title: Sleep Intervention for Youth With Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Responsible Party: Principal Investigator, Michelle Perfect, Associate Professor, University of Arizona
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 12-0733091
Record Dates: First submitted 2012-11-29; First posted 2012-12-03 (Estimated); Last update posted 2016-11-21 (Estimated); Status verified 2016-11

CONDITIONS: Diabetes
Keywords: Diabetes; Sleep problems; School; Neurobehavioral
MeSH Terms: conditions — Diabetes Mellitus; Parasomnias

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sleep Extension (Experimental): All youth in this condition are asked to extend their sleep to 10 hours or at least one hour, whichever is longer
  Interventions: Behavioral: Sleep extension
- Fixed Sleep Duration (Sham Comparator): All youth in this condition are asked to maintain their baseline sleep duration.
  Interventions: Behavioral: Fixed Sleep Duration

INTERVENTIONS:
Behavioral: Sleep extension — There will be a consultation with families to help youth to be successful in extending their sleep.
  Arms: Sleep Extension
Behavioral: Fixed Sleep Duration — There will be a consultation with families to instruct youth to maintain the same average nightly sleep duration during the modification week. The purpose is to control for time and attention.
  Arms: Fixed Sleep Duration

SUMMARY:
Sleep intervention for youth with diabetes

DETAILED DESCRIPTION:
It is known that sleep disturbances in healthy youth have negative effects on neurobehavioral functioning. Further, data support that individuals with diabetes have more sleep disturbances and compromised neurobehavioral functioning than individuals without diabetes. However, the joint impact of sleep and glucose on neurobehavioral functioning in youth with type 1 diabetes (T1DM) is not yet known. Therefore, our primary study aims are to: (1) determine the relative contributions of various sleep disturbances on glucose control in youth with T1DM; (2) examine the joint impact of glucose control and sleep disturbances on neurobehavioral outcomes in youth with T1DM; and (3) determine if increasing sleep duration relative to youth's typical schedules contributes to changes in glycemic control and neurobehavioral performance. These aims will be achieved by following 120 youth with T1DM ages 10 through 16 for six days of naturalistic sleep using polysomnography, actigraphy, and questionnaires to assess sleep; continuous glucose monitors and hemoglobin A1C values to assess glucose control; and standardized cognitive tasks and behavior rating scales to assess neurobehavioral functioning. Further, the proposed study is innovative in that it will extend existing research by moving from correlational findings to an experimental paradigm by randomizing youth with T1DM to either a Sleep Extension or Fixed Sleep Duration condition for an additional six days. Once our aims are achieved and a causal link is established, the proposed Sleep Extension intervention will advance knowledge about the role of sleep in diabetes management and provide a beneficial intervention to help youth with T1DM.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of type 1 diabetes
* enrolled in school

Exclusion Criteria:

* not hospitalized within past month
* neurological, developmental, or psychiatric condition that in the opinion of the PI would significantly interfere with sleep or participation

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 114 (Actual)
Dates: Start 2012-10; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Academic Rating Scale | 2 weeks
  A teacher behavioral rating of classroom behaviors and performance
Glucose control | 2 weeks
  Continuous glucose monitor
Neurocognitive performance | 2 weeks
  Cogstate learning and memory tasks
Academic performance | 2 weeks
  Woodcock Johnson Tests of Achievement-3rd Edition NU and Curriculum-Based Measurements

CONTACTS AND LOCATIONS:
Overall Officials: Michelle M Perfect, PhD, Principal Investigator — UA College of Education
Locations (1):
- Angel Wing Clinic for Diabetes, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
Upon request.